CLINICAL TRIAL: NCT06747975
Title: Preventative Effect of Combining Dexamethasone with Ondansetron on Postoperative Nausea, Vomiting and Shivering in Children Undergoing Caudal Anesthesia
Brief Title: Preventative Effect of Combining Dexamethasone with Ondansetron on Postoperative Nausea, Vomiting and Shivering in Children Undergoing Caudal Anesthesia on Hypospadias Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Fathy Ahmed, resident doctor at Assiut University hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dexamethasone+ondansetron PONV
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Caudal Anesthesia
Keywords: dexamethasone; ondansetron
MeSH Terms: interventions — Dexamethasone; Ondansetron; Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group A (Experimental): fifty patients will receive Caudal epidural block (0.5 mL/kg of bupivacaine 0.25% plus dexa- methasone 0.1 mg/kg plus 4mg ondansetron ), and IV 5 mL normal saline
  Interventions: Drug: Dexamethasone and Ondansetron; Drug: Bupivacaine + saline
- group B (Placebo Comparator): fifty patients will receive Caudal epidural block (0.5 mL/kg of bupivacaine 0.25% plus dexa- methasone 0.1 mg/kg plus 4mg ondansetron ), and IV 5 mL normal saline
  Interventions: Drug: Bupivacaine + saline

INTERVENTIONS:
Drug: Dexamethasone and Ondansetron — patients will receive Caudal epidural block (0.5 mL/kg of bupivacaine 0.25% plus dexa- methasone 0.1 mg/kg plus 4mg ondansetron ), and IV 5 mL normal saline
  Arms: group A
Drug: Bupivacaine + saline — patients will receive caudal epidural block (0.5 mL/kg of bupivacaine 0.25% only) and IV 5 mL normal saline

SUMMARY:
caudal epidural block is a technique used as an adjuvant to general anesthesia for postoperative analgesia in pediatric patients,especially those with infraumbilical, perineal and lower extremity surgery , because it reduces the need for perioperative and postoperative analgesia, reduces the need for general anesthesia, accelerates the awakening, suppresses the surgical neurohumoral stress response and can be performed easily The objective of the current study is to determine the efficacy and safety of prophylactic intravenous administration of combination of 0.1mg/kg of dexamethasone plus 4mg of ondansetron immediately before establishment of caudal block for prevention of Nausea&vomiting and Shivering in pediatric patients undergoing infra umbilical surgeries

DETAILED DESCRIPTION:
Although it has some adverse effects: postoperative nausea and vomiting (PONV) are frequent and morbidity-related complication in children, PONV is still present in almost twice the frequency of adults, 33.2-82%. shivering is one of frequent, undesirable adverse effects, The incidence of shivering is up to 40-60% even in regional anaesthesia leads to O2 consumption and CO2 production,So we target in this study two effective drugs with less side effects to reduse these adverse effects Ondansetron is a highly potent selective 5 hydroxytryptamine receptor antagonist, which is widely used as an anti-emetic, Its mechanism of action as anti-shivering is not clear and it is proposed to act centrally at the level of the pre-optic anterior hypothalamic region by inhibition of serotonin reuptake Dexamethasone: is a potent class of steroid drugs ,It prevents thermoregulatory shivering via its central inhibitory effect on the thermoregulatory center and prevents non thermoregulatory shivering by its anti-inflammatory activity, i.e. antagonizing the activation of the inflammatory responses and release of cytokines during surgery The anti-emetic properties of dexamethasone are well established but the mechanisms underlying this anti-emetic effect remain largely unknown

ELIGIBILITY:
Inclusion Criteria: -

* Age from 2 to 12 years old.
* Patients with stable vital signs.
* Patients with normal laboratory investigations.
* Patients undergoing Caudal anaesthesia for infraumbilical surgeries

Exclusion Criteria: -

* Patient's parental refusal.
* Age < 2 or > 12 years.
* Contraindications to Caudal anaesthesia (Coagulopathy, increased intracranial pressure, or local skin infection ,pilonidal cyst and congenital anomalies of lower spine because of unclear or impalpable anatomy
* Patients with cardiac morbidities.
* Failure of caudal block
* Diabetes mellitus
* Convulsions.
* Known allergy to any drugs used in this study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of all emesis | 24 hours
  the incidence of all emesis in the 24 h after surgery (PONV).

IPD SHARING:
Plan to Share IPD: Undecided